CLINICAL TRIAL: NCT03489746
Title: A Cluster Randomised Trial of Medication Review and Withdrawal of Inappropriate Inhaled Corticosteroid Treatment in Chronic Obstructive Pulmonary Disease
Brief Title: Steroid Withdrawal Intervention in Fife and Tayside
Acronym: SWIFT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely but potentially will resume
Sponsor: NHS Tayside (Other Government)
Collaborators: NHS Fife (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016RC23
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inhaled corticosteroids; Quality improvement; Cluster randomized Trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial at practice level
Who Masked: Investigator, Outcomes Assessor
Masking Description: All data will be analysed anonymously
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled corticosteroid withdrawal (Experimental): Patients meeting the study criteria for withdrawal will have their ICS containing regime changed to a LABA/LAMA regime without ICS.
  Interventions: Other: ICS withdrawal protocol
- Standard care (Active Comparator): Patients will continue on their current recommended regimen including ICS.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: ICS withdrawal protocol — A primary care intervention to support switch from ICS containing regimen to non-ICS containing regimen in appropriate patients.
  Arms: Inhaled corticosteroid withdrawal
Other: Standard care — Normal clinically indicated inhaled therapy
  Arms: Standard care

SUMMARY:
The SWIFT trial is a cluster randomised trial to determine if a patient identification, feedback and inhaled corticosteroid (ICS) withdrawal intervention in primary care can result in more appropriate inhaled corticosteroid use without increasing the frequency of exacerbations. Practices in Tayside and Fife will be randomised at practice level to an intervention or control. The intervention will consist of electronic review of patients Chronic obstructive pulmonary disease (COPD) data and prescribing history, followed by implementation of a medication change involving withdrawal of ICS and introduction of a Long acting beta adrenergic agonist (LABA) and Long acting muscarinic antagonist (LAMA) for patients without an indication for ongoing ICS treatment. Patients in control practices will not receive the intervention, but practices will be provided with local guidelines and formulary and encouraged to prescribe appropriately. Patients in the control practices may be switched to guideline compliant medications. Our hypothesis is that removal of non-evidence barriers to appropriate prescribing will result in in high rates of ICS withdrawal and that the intervention will be safe, as evidenced by no increase in the frequency of exacerbations over 12 months of follow-up.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide and a major cause of morbidity in the UK. Inhaled corticosteroids (ICS) are frequently prescribed to patients with COPD and these medications represent a major burden on the National Health Service in terms of drug costs. They are not without side effects, and pneumonia in particularly has been highlighted as a common adverse event in COPD patients receiving ICS.

In the UK, inhaled corticosteroids are indicated for patients with severe or very severe COPD (Forced expiratory volume in 1 second <50% predicted) who experience frequent exacerbations. International guidelines and strategies such as those from Global Obstructive Lung Disease (GOLD), also suggest inhaled corticosteroids should be reserved for patients with frequent exacerbations despite appropriate treatment with inhaled bronchodilators such as combined long acting beta-agonists and long acting muscarinic antagonists (LABA/LAMA combinations). Despite this guidance, use of inhaled corticosteroids in patients with milder COPD and without a history of exacerbations is common. Randomised controlled trials suggest that inhaled corticosteroids can be withdrawn from COPD patients with minimal adverse effects. Attempts to reduce inappropriate ICS prescribing have been largely unsuccessful in real-life, however, because of "non-evidence barriers". These include a lack of expertise in general practice to identify patients suitable for ICS withdrawal, fear of adrenal insufficiency, concern about missing a diagnosis of asthma and time. A high proportion of COPD care in the United Kingdom is delivered by specialist practice nurses, who may not be empowered to withdraw ICS in the absence of specific guidance or protocols.

The SWIFT trial is a cluster randomised trial to determine if a patient identification, feedback and ICS withdrawal intervention in primary care can result in more appropriate inhaled corticosteroid use without increasing the frequency of exacerbations. Practices in Tayside and Fife will be randomised at practice level to an intervention or control. The intervention will consist of electronic review of patients COPD data and prescribing history, followed by implementation of a medication change involving withdrawal of ICS and introduction of a LABA/LAMA for patients without an indication for ongoing ICS treatment. Patients in control practices will not receive the intervention, but practices will be provided with local guidelines and formulary and encouraged to prescribe appropriately. Patients in the control practices may be switched to guideline compliant medications (which may include the withdrawal of inhaled corticosteroids).

Our hypothesis is that the above "non-evidence barriers" will result in an ongoing high inappropriate use of ICS in control practices while an intervention that overcomes these will result in high rates of ICS withdrawal and that the intervention will be safe, as evidenced by no increase in the frequency of exacerbations over 12 months of follow-up.

This study will make an important contribution to understanding the role of inhaled corticosteroids in COPD. If successful, the intervention could be safely applied throughout the NHS to reduce inappropriate medication use, reduce patient side effects and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged > 40 years
* A clinical diagnosis of COPD made by a physician
* Post-bronchodilator FEV1/FVC ratio at screening of <70%

Exclusion Criteria:

* Asthma recorded in general practice records or clinically suspected
* Patients with COPD receiving inhaled short acting beta-2 agonist only.
* Residence outwith Tayside and Fife
* Insufficient data available to determine appropriateness of ICS and other medication use.
* Known previous failure of inhaled corticosteroid withdrawal
* Patients should be excluded if, in the opinion of the practice, making changes to their current COPD treatment regime is not in the patients best interests.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of moderate and severe exacerbations of COPD | 1 year
  Use of corticosteroids and/or antibiotics (moderate) or hospitalization (severe) for exacerbation of COPD

SECONDARY OUTCOMES:
Respiratory Hospitalizations | 1 year
Success of ICS withdrawal | 1 year
  Inhaled corticosteroid prescribing rates (number of patients receiving inhaled corticosteroid prescriptions at study completion divided by total number of COPD patients) and withdrawal rates (number of patients receiving inhaled corticosteroids prior to the intervention divided by the number of patients receiving inhaled corticosteroids following the intervention in each arm)
Time to the first moderate and severe exacerbation | Time to first event (patients without an event censored at 1 year)
  First exacerbation or respiratory hospitalisation following the intervention
Oral corticosteroid use | 1 year
  Cumulative prescriptions for oral corticosteroids (excluding chronic low dose oral corticosteroids)
Antibiotic use | 1 year
  Cumulative prescriptions for oral antibiotics (excluding chronic low dose macrolides)

OTHER OUTCOMES:
Rates of known ICS related adverse effects between groups | 1 year
  Pneumonia, fractures, cataracts and diabetes
Rates of ICS relapse | 1 year
  Proportion of patients undergoing ICS withdrawal who are subsequently restarted on inhaled corticosteroids within 12 months
Mortality | 1 year
  GRO based mortality data
Subgroup analyses in patients successfully withdrawing ICS | 1 year
  Frequency of moderate and severe exacerbations
Subgroup analyses based on baseline lung function for major endpoints | 1 year
  Frequency of moderate and severe exacerbations
Subgroup analyses based on baseline eosinophil count <300 cells/ul for major endpoints | 1 year
  Frequency of moderate and severe exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Short, Principal Investigator — NHS Tayside; Devesh Dhasmana, Principal Investigator — NHS Fife; Arlene Shaw, Study Director — NHS Tayside; Fiona Eastop, Study Director — NHS Tayside
Locations (2):
- United Kingdom (2):
  - NHS Tayside, Dundee, Perthshire
  - NHS FIfe, Kirkcaldy

IPD SHARING:
Plan to Share IPD: Yes
Data will be publically available through the health informatics centre, University o fDundee
Supporting Information: Study Protocol, SAP
Time Frame: To be determined
Access Criteria: Open